CLINICAL TRIAL: NCT02593097
Title: Metformin for the Prevention of Episodic Migraine: a Randomized, Double-blind, Placebo-controlled, Crossover Study
Brief Title: Metformin for the Prevention of Episodic Migraine (MPEM)
Acronym: MPEM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Amaal J. Starling, M.D., Assistant Professor, Mayo Clinic
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 15-000422
Record Dates: First submitted 2015-10-28; First posted 2015-10-30 (Estimated); Results first posted 2020-07-01 (Actual); Last update posted 2020-07-01 (Actual); Status verified 2020-06

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Metformin first, then matching placebo (Experimental): Subjects will be randomized into the Metformin group, treated for 12 weeks with a 4 week washout period in between treatments, then treated with matching placebo for 12 weeks.
  Interventions: Drug: Metformin; Drug: Matching Placebo
- Matching placebo first, then Metformin (Experimental): Subjects will be randomized into the matching placebo group, treated for 12 weeks with a 4 week washout period in between treatments, then treated with Metformin for 12 weeks.
  Interventions: Drug: Metformin; Drug: Matching Placebo

INTERVENTIONS:
Drug: Metformin — Metformin 500mg twice daily
Drug: Matching Placebo — Matching Placebo twice daily
  Other Names: Placebo

SUMMARY:
The investigators will evaluate the safety and efficacy of metformin for preventive treatment of migraine in a randomized, double-blind, placebo-controlled, crossover trial.

DETAILED DESCRIPTION:
This will be a single-center, double-blind, randomized, placebo-controlled, crossover study. The investigators will enroll 40 subjects. Subjects will be recruited from the outpatient Mayo Headache Clinic, Mayo Women's Health Clinic, Mayo Community Internal Medicine, and the Mayo Clinic- Arizona State University Neurology Clinic. The Headache Clinic employs 6 headache specialists and 1 fellow which is sufficient staffing to support this study and recruitment of patients with migraine.

Before study enrollment, patients will undergo a 2-hour oral glucose tolerance test to confirm the absence of diabetes mellitus.

Subjects will then keep a headache diary for 4 weeks to establish baseline characteristics, including number of migraine days per month, number of moderate to severe headache days per month, and number of days per month of acute medication use. The 4-week baseline period will be followed by 2 treatment periods of 12 weeks each, separated by a washout period of 4 weeks (total study duration, 32 weeks). For the 12-week treatment periods, subjects will receive either metformin 500mg twice daily or matching placebo twice daily.

Subjects will have 7 study visits. Routine laboratory studies and a pregnancy test will be performed at enrollment and week 20. Abnormal kidney or liver function will exclude subjects. Pregnancy will exclude subjects. General and neurologic examinations will be performed during 3 of the 7 visits. At each visit, subjects will receive medication for the period until the next visit. A headache diary will be used for the trial. For every day that the subject has a headache of any type, she or he will record headache characteristics, associated features, and medications used.

ELIGIBILITY:
Inclusion Criteria:

1. age 18-65 years
2. a diagnosis of migraine with or without aura for >1 year according to the International Classification of Headache Disorders-IIIb

Exclusion Criteria:

1. a diagnosis of diabetes mellitus or polycystic ovarian syndrome
2. overuse of acute migraine treatments
3. failure to respond to 3 or more classes of preventive drug treatments
4. change in dose of migraine-preventive medication within 2 months of beginning the baseline diary phase
5. significant somatic or psychiatric disease
6. known alcohol or other substance abuse
7. pregnant or breastfeeding.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2016-02; Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amaal J Starling, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Price TJ, Dussor G. AMPK: An emerging target for modification of injury-induced pain plasticity. Neurosci Lett. 2013 Dec 17;557 Pt A(0 0):9-18. doi: 10.1016/j.neulet.2013.06.060. Epub 2013 Jul 3. PMID 23831352
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Metformin First, Then Matching Placebo: Subjects who received Metformin in either the first or last 12 weeks of the study
  Subjects will be randomized into the Metformin group, treated for 12 weeks with a 4 week washout period in between treatments, then treated with matching placebo for 12 weeks.
  Metformin: Metformin 500mg twice daily
  Matching Placebo: Matching Placebo twice daily
- Matching Placebo First, Then Metformin: Subjects who received matching placebo either the first or last 12 weeks of the study
  Subjects will be randomized into the matching placebo group, treated for 12 weeks with a 4 week washout period in between treatments, then treated with Metformin for 12 weeks.
  Metformin: Metformin 500mg twice daily
  Matching Placebo: Matching Placebo twice daily
Period: First Intervention (12 Weeks)
Arm/Group | Metformin First, Then Matching Placebo | Matching Placebo First, Then Metformin
Started | 14 | 20
Received Intervention | 14 | 20
Completed | 12 | 16
Not Completed | 2 | 4
Not completed — Lost to Follow-up | 1 | 2
Not completed — Withdrawal by Subject | 1 | 2
Period: Washout (4 Weeks)
Arm/Group | Metformin First, Then Matching Placebo | Matching Placebo First, Then Metformin
Started | 12 | 16
Completed | 12 | 16
Not Completed | 0 | 0
Period: Second Intervention (12 Weeks)
Arm/Group | Metformin First, Then Matching Placebo | Matching Placebo First, Then Metformin
Started | 12 | 16
Completed | 9 | 15
Not Completed | 3 | 1
Not completed — Lost to Follow-up | 1 | 1
Not completed — Lack of Efficacy | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Metformin First, Then Matching Placebo | Matching Placebo First, Then Metformin | Total
Number analyzed (Participants) | 14 | 20 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.85 (6.91) | 46.83 (10.94) | 45.34 (8.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 17 | 28
  Male | 3 | 3 | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 14 | 20 | 34

OUTCOME MEASURES:

1. Primary Outcome: Headache Days
Description: Total number of moderate and severe headache days
Time Frame: Baseline through end of study for a total of approximately 32 weeks
Population: Data was only analyzed for the subjects that completed both interventions.
Measure: Mean (Standard Deviation); unit: Days
Groups:
- Metformin: Subjects who received Metformin in either the first or last 12 weeks of the study
- Matching Placebo: Subjects who received matching placebo either the first or last 12 weeks of the study
Arm/Group | Metformin | Matching Placebo
Number analyzed (Participants) | 30 | 32
Days | 23.64 (2.15) | 24.33 (2.19)
Statistical Analysis 1: Comparison: Metformin vs Matching Placebo; Test type: Superiority; p = 0.83, Hills-Armitage

2. Secondary Outcome: Greater Than >50% Reduction in Migraine Days on Metformin
Description: Percentage of patients whose migraines reduced by at least 50% on Metformin.
Time Frame: 12 weeks
Population: Data was not collected for the matching placebo arm. This outcome measure was specific for metformin, no analysis was done for the placebo.
Measure: Mean (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Metformin | Matching Placebo
Number analyzed (Participants) | 30 | 0
percentage of subjects | 10.1 [-3.46 to 23.66] |
Statistical Analysis 1: Comparison: Metformin; Test type: Superiority; p = 0.16, McNemar

3. Secondary Outcome: Adverse Events
Description: Total number of subjects with treatment-related adverse events
Time Frame: Baseline through end of study for a total of approximately 32 weeks
Population: Data was only analyzed for the subjects that completed both interventions.
Measure: Count of Participants; unit: Participants
Arm/Group | Metformin | Matching Placebo
Number analyzed (Participants) | 30 | 32
Participants | 3 | 1

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from a period of baseline to four weeks post last intervention for a total of approximately 32 weeks
Description: Safety population included all participants who received at least one dose of intervention.
Arm/Group | Metformin | Matching Placebo
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/32
Other Adverse Events (participants affected / at risk) | 12/30 | 4/32
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metformin (N=30) | Matching Placebo (N=32)
Dry Mouth (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 1 (1)
Dry hair (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
Hair loss (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-12): https://cdn.clinicaltrials.gov/large-docs/97/NCT02593097/Prot_SAP_000.pdf